CLINICAL TRIAL: NCT04432662
Title: Darbepoetin in Neonatal Encephalopathy (EDEN) Trial
Brief Title: Darbepoetin in Neonatal Encephalopathy Trial
Acronym: EDEN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 277361
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Neonatal Encephalopathy
MeSH Terms: interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Darbepoetin Alpha (Active Comparator): Administration of Darbepoetin Alpha (10 mcg/kg) IV x2 doses following cooling therapy.
  Interventions: Drug: Darbepoetin Alfa
- Standard of care (No Intervention): Standard of care: Cooling only

INTERVENTIONS:
Drug: Darbepoetin Alfa — Administration of Darbepoetin Alpha (10 mcg/kg) IV x2 doses following cooling therapy.
  Arms: Darbepoetin Alpha

SUMMARY:
Hypoxic Ischemic Encephalopathy is also known as 'birth asphyxia related brain injury' and happens when the brain does not receive enough oxygen or blood flow around the time of birth. Birth asphyxia related brain injury is the most common cause of death and neurodisability in term babies.

Cooling therapy has substantially improved the outcomes of babies with HIE. However, unacceptably high rate of adverse outcomes are still seen in cooled babies with HIE.

The EDEN trial is a 2 arm randomised control trial and aims to examine the physiological effects of Darbepoetin alfa (Darbe) therapy on proton magnetic resonance spectroscopy thalamic N-acetylaspartate (NAA) level in babies with neonatal encephalopathy undergoing cooling therapy.

A total of 150 babies with neonatal encephalopathy will be recruited from the participating sites in UK over a 24 month period. The babies will be randomly allocated to darbepoetin or usual care. MR imaging and spectroscopy will be performed at 1 to 2 weeks of age to examine the brain injury. Neurodevelopmental outcomes will be assessed at 18 months of age.

DETAILED DESCRIPTION:
Birth asphyxia related brain injury occurs in 2.6 (95% CI 2.5 to 2.8) per 1000 live births in the UK and is the most common cause of death and neurodisability in term babies. The economic burden to the treasury on support costs of neurodisability from neonatal encephalopathy is massive (£4 billion per year). In addition, birth asphyxia related (obstetric) claims accounted for almost half of the NHS litigation expenses in 2016/17 (approx. £2 billion), increasing by 15% from the previous year. It has been reported that the NHS cost to meet the complex life-long care needs of babies born with brain damage could be soon over £20m per child, and this situation is unsustainable to the NHS.The UK Government has recently (October 2016) announced that reducing birth asphyxia related costs is a priority area for the Government.

The only effective treatment for neonatal encephalopathy is whole-body cooling, with an estimated saving of £100 million per annum to the UK economy, since its introduction as standard therapy in the NHS in 2007. Cooling therapy has substantially improved the outcomes of babies with neonatal encephalopathy in the past decade. However, unacceptably high rate of adverse outcomes are still seen in cooled babies with moderate or severe neonatal encephalopathy : death 28% (range 24-38); cognitive impairment 24% (range 21-25); cerebral palsy 22% (range 13-28); epilepsy 19% (range 15-24); cortical visual impairment 6% (range 1-10), with combined death or moderate/severe disability 48% (range 44- 53), and hence better treatments and further optimisation of cooling therapy is required. Additionally, cooling provides a window of opportunity for therapeutic interventions that may arrest or reduce secondary brain injury and it is unclear whether it provides protection from a sub-acute chronic injury that may have occurred during the antenatal period.

A key roadblock in clinical translation of over fifteen highly effective neuroprotective treatments in animal models is the long delay between the intervention and outcome assessments in neonatal encephalopathy . i.e., the earliest age at which neurodevelopmental outcome can be accurately assessed is 18 months. Hence, despite having several highly effective treatments in animal models, no further neuroprotective drugs in neonatal encephalopathy have been introduced into the NHS in the past ten years.

Erythropoietin (Epo) is a widely used drug for treating anaemia in various age groups, including newborn infants. Several recent reviews have highlighted Epo as one of the most promising therapies to augment hypothermic neuroprotection. Epo has both acute effects (anti-inflammatory, anti-excitotoxic, anti-oxidant, and anti-apoptotic) and regenerative effects (neurogenesis, angiogenesis, and oligodendrogenesis) essential for the repair of injury and normal neurodevelopment in animal models. Of the long list of highly effective drugs in animal models of neonatal encephalopathy and early clinical studies, Epo is the most promising. It is the only drug with a long therapeutic window, is widely available, inexpensive, and can be easily administered on a once-a-day dosing schedule. It has been extensively evaluated in large randomised controlled trials for anaemia of prematurity and has a proven safety profile in newborn infants. Due to the regenerative effects and the longer therapeutic window provided by Epo, there is potential to impact the chronic injury caused to an antenatally compromised foetus.

Although earlier studies have shown benefit with Epo, the time of initiation and duration of treatment remains uncertain. Moreover, recently published High-Dose Erythropoietin for Asphyxia and Encephalopathy (HEAL) trial which administered high dose Epo (1000u/kg/day) within 24 hours of birth and continued until 7 days of age failed to demonstrate the neuroprotective effect of erythropoietin in moderate and severe encephalopathy as an adjuvant to therapeutic hypothermia. This result suggest the exposure of the drug during the therapeutic hypothermia may not be beneficial due to an overlap in the neuroprotective mechanism. Perhaps a prolonged exposure of Epo following therapeutic hypothermia might be beneficial.

Another erythropoiesis stimulating agent is Darbepoetin (Darbe) with dual erythropoietic and potential neuroprotective effects. Darbe is an ideal candidate to augment hypothermic neuroprotection as it is a long-acting erythropoiesis stimulating agent, allowing prolonged exposure with less dosing. In preclinical study in rats, darbepoetin alfa crossed the blood brain barrier and remained stable up to 24 hours. Neuroprotective effects of darbepoetin were demonstrated following the contusion injury and hemorrhage in rats. The DANCE study (Darbepoetin Administered to Neonates undergoing Cooling for Encephalopathy) randomised 30 term infants with moderate to severe neonatal encephalopathy to placebo (n=10), 2 μg/kg Darbe (n=10) or 10 μg/kg Darbe (n=10). At 2 and 10 μg/kg Darbe, t1/2 was 24 and 32 hours. A dose of 10 μg/kg dose achieved an AUC in the neuroprotective range and a terminal t1/2 of 53.4 hours when compared to the 2 μg/kg dose. No side effects attributable to Darbe were reported. In another feasibility and safety trial, infants with mild encephalopathy were randomised to receive Darbepoetin 10 μg/kg single dose within 24 hours and found the drug to be safe with no reported adverse events.

The EDEN trial is a 2 arm randomised control trial and aims to examine the physiological effects of Darbepoetin alfa (Darbe) therapy on proton magnetic resonance spectroscopy thalamic N-acetylaspartate (NAA) level in babies with neonatal encephalopathy undergoing cooling therapy.

After informed parental consent, a total of 150 babies with HIE (aged <24 hours) undergoing therapeutic hypothermia will be randomised to one of the following groups

* Arm 1:Darbepoetin Alpha (10 mcg/kg) IV x2 doses following cooling therapy.
* Arm 2: Cooling only (usual care)

Babies recruited will have electroencephalography (EEG), MR imaging and spectroscopy will be performed at 1 to 2 weeks of age to examine the brain injury. The neurological outcomes will be assessed between 18 to 22 months of age. The trial duration will be 4 years, consisting of a 4 week start up period, 24 month recruitment period, a 18 month follow-up period, and 5 months for data analysis and write up.

ELIGIBILITY:
Inclusion Criteria:

All the following criteria should be met

1. Babies aged < 24 hours, gestation age >36 weeks with a birthweight >1.8kg.
2. Acute perinatal asphyxia (metabolic acidosis in cord and/or blood gas (pH<7.0; base deficit > 16 mmol/L) within first 1 hour of birth). If pH between 7.01 and 7.15, a base deficit between 10 and 15.9 mmol/L, additionally acute obstetric event and either need for continued resuscitation or ventilation at 10 minutes after birth and/or 10 minutes Apgar score <5 is required.
3. Evidence of mild, moderate, or severe encephalopathy on an NICHD neurological examination performed between 1 and 6 hours of birth. The worst recorded encephalopathy stage between 1 and 6 hours of birth should be used.
4. Cooling therapy initiated for neonatal encephalopathy within 6 hours of age as a part of standard clinical care, with an intention of continuing for 72 hours.

Exclusion Criteria:

1. Major life-threatening congenital malformation.
2. Concomitant participation in other research projects

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure (Mean (SD) of thalamic NAA level) | Expected average 1 to 2 weeks after birth
  Mean (SD) of thalamic NAA level in babies treated with Darbe when compared with untreated infants.

SECONDARY OUTCOMES:
Secondary outcome measure (accurate quantification of NAA level) | 24 months
  Number of babies in whom thalamic NAA level could be accurately quantified in 3Telsa and 1.5Tesla MR scanners.

CONTACTS AND LOCATIONS:
Locations (9):
- United Kingdom (9):
  - Birmingham Womens Hospital, Birmingham
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Medway NHS Foundation Trust, Gillingham
  - Liverpool Womens NHS Foundation Trust, Liverpool
  - Homerton University Hospital, London
  - Imperial College Healthcare Trust, London
  - Bedfordshire Hospitals NHS Foundation Trust, Luton
  - The Newcastle Upon Tyne NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: Yes
IPD data will be shared for meta-analysis
Supporting Information: Study Protocol, ICF
Time Frame: 2 years after the trial is published
Access Criteria: Quality of the meta-analysis and the credibility of the team

REFERENCES:
- [Background] Lally PJ, Montaldo P, Oliveira V, Soe A, Swamy R, Bassett P, Mendoza J, Atreja G, Kariholu U, Pattnayak S, Sashikumar P, Harizaj H, Mitchell M, Ganesh V, Harigopal S, Dixon J, English P, Clarke P, Muthukumar P, Satodia P, Wayte S, Abernethy LJ, Yajamanyam K, Bainbridge A, Price D, Huertas A, Sharp DJ, Kalra V, Chawla S, Shankaran S, Thayyil S; MARBLE consortium. Magnetic resonance spectroscopy assessment of brain injury after moderate hypothermia in neonatal encephalopathy: a prospective multicentre cohort study. Lancet Neurol. 2019 Jan;18(1):35-45. doi: 10.1016/S1474-4422(18)30325-9. Epub 2018 Nov 15. PMID 30447969